CLINICAL TRIAL: NCT03813680
Title: Comparison Between Passive Vertebral Mobilization and Proprioceptive Neuromuscular Techniques in Managing Pain and Disability in Patients With Mechanical Neck Pain
Brief Title: Passive Vertebral Mobilization and Propriocemptive Neuromuscular Techniques in Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Muhammad Ashfaq, Principal Investigator, Isra University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1402-PhD-003
Record Dates: First submitted 2019-01-13; First posted 2019-01-23 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Mechanical Neck Pain
Keywords: Mechanical Neck Pain; Passive Vertebral Mobilization; Proprioceptive Neuromuscular Techniques (PNF); Quality of Life; Disability; Pain
MeSH Terms: conditions — Pain | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PVM group (Active Comparator): This group included 30 participants. Passive vertebral mobilization was given along with routine physiotherapy comprising TENS, Hotpack/IRR, Isometric neck exercise and postural care
  Interventions: Other: Passive Vertebral Mobilization; Other: Routine Physiotherapy
- PNF group (Active Comparator): This group included 30 participants. PNF exercise in the form of diagonal pattern neck movements was along with routine physiotherapy comprising TENS, Hotpack/IRR, Isometric neck exercise and postural care
  Interventions: Other: PNF exercise; Other: Routine Physiotherapy
- RPT(Routine Physiotherapy) group (Active Comparator): This group included 30 participants.Routine physiotherapy comprising TENS, Hotpack/IRR, Isometric neck exercise and postural care.
  Interventions: Other: Routine Physiotherapy

INTERVENTIONS:
Other: Passive Vertebral Mobilization — Posteroanterior glides was given to cervical spine using Maitland method along with routine physiotherapy comprising thermotherapy with Hot Packs 15 minutes, Transcutaneous Electrical Nerve Stimulation (TENS) 15 minutes,Isometric neck exercises,Education on precautions and postural care
  Other Names: Spinal mobilization
  Arms: PVM group
Other: PNF exercise — The subjects was given PNF exercises comprising PNF diagonal patterns for neck along with routine physiotherapy comprising thermotherapy with Hot Packs 15 minutes, Transcutaneous Electrical Nerve Stimulation (TENS) 15 minutes,Isometric neck exercises,Education on precautions and postural care
  Other Names: Proprioceptive Neuromuscular Facilitation
  Arms: PNF group
Other: Routine Physiotherapy — Thermotherapy with Hot Packs 15 minutes, Transcutaneous Electrical Nerve Stimulation (TENS) 15 minutes,Isometric neck exercises,Education on precautions and postural care
  Other Names: Routine Physical therapy (RPT)

SUMMARY:
This study was conducted to determine the effectiveness of Passive Vertebral Mobilization (PVM) and Proprioceptive Neuromuscular Techniques (PNF) in reducing pain, disability and improving quality of life in patients with Mechanical Neck Pain.

DETAILED DESCRIPTION:
Neck Pain is very common and is now considered a public health issue. It poses significant health and economic burden, being a frequent cause of disability. A significant proportion of direct health care costs associated with neck disorders are attributable to visits to health care providers, to sick leave, and to the related loss of productive capacity. Mechanical neck pain affects between 45-54% of people in the general population .This can result in severe pain and disability. Mechanical neck pain described as a reduction in the mobility of cervical spinal segment is often the focus of manipulative physical therapy interventions. Most neck pain is not attributed to diseases but rather caused by muscular and postural condition. The cervical pain is a mechanical problem .It is therefore sense that a mechanical treatment works better than pharmacological treatment.

Cervical spine often impairs flexibility of key muscles related to cervical spine . Stretching exercise is beneficial for increasing flexibility as well as muscle performance.

The normal function of cervical spine is complex and requires a large variety of activities to be coordinated in order for an individual to perform daily activities with the least amount of strain and potential injury. When the dysfunction develops in the cervical spine, a chain reaction may develop which can affect the whole neck and even the entire body.

Commonly used approaches to treatment include rest, therapeutic massage, application of physical agents like heat, cold, TENS, and ultrasonic various types of mobilizations, manipulations (by physical therapists, chiropractors, osteopaths and others), therapeutic exercises, postural care and off course medication and surgical interventions. However, studies of their effectiveness have generally been short-term and inconclusive. The aim of the study is to compare which treatment either Passive Vertebral Mobilization or Proprioceptive Neuromuscular Facilitation, whether itself or in combination, is more effective and beneficial in the treatment of mechanical neck pain.

Several studies have been reported to determine the effectiveness of manual therapy/ passive vertebral mobilization but with largely inconclusive results. However there are few studies if any to compare PNF exercise with PVM in terms of their effectiveness. PNF are simple and requiring low level expertise as compare to PVM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mechanical neck pain having limited range of motion and muscle spasm and difficulty function between 18 to 60 years of age

Exclusion Criteria:

* Patients diagnosed with rheumatoid arthritis, Ankylosing spondylitis or other systemic disease
* Patients with cancer of the cervical spine
* Patients with history of fracture of spine
* Patients with any congenital anomaly of Cervical spine
* Patients having whiplash disorder with in last four weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-09-20 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (PAIN) | 4 weeks
  changes from baseline. Visual Analog Scale (VAS) is a 10 cm horizontal line, with 0 presenting No pain and 10 representing Worst Pain.
ROM of Cervical spine (Flexion) | 4 weeks
  changes from baseline
ROM of Cervical spine (Extension) | 4 weeks
  changes from baseline.Bubble inclinometer was used to measure ROM in sitting position
ROM of Cervical spine (rotation rightward) | 4 weeks
  changes from baseline.Bubble inclinometer was used to measure ROM in sitting position
ROM of Cervical spine (rotation leftward) | 4 weeks
  changes from baseline. Bubble inclinometer was used to measure ROM in sitting position
ROM of Cervical spine (Side bending Right) | 4 weeks
  changes from baseline.Bubble inclinometer was used to measure ROM in sitting position
ROM of Cervical spine (Side bending Left) | 4 weeks
  changes from baseline.Bubble inclinometer was used to measure ROM in sitting position
Neck Flexors Muscle endurance | 4 weeks
  changes from baseline. Neck Flexion holding time in supine lying position was measured in seconds with the help of stop watch.
NDI (neck Disability Index) | 4 weeks
  changes from baseline NDI is self rated index to measure pain and disability due to neck pain.
  Neck disability index consists of 10 questions addressing functional activities. There are 6 potential responses for each item, ranging from no disability (0) to total disability (5).The NDI is scored from 0 to 50 with higher score indication greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ashfaq, Principal Investigator — Isra University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashfaq M, Babur MN, Malick WH, Hussain MA, Awan WA. Comparative effectiveness of proprioceptive neuromuscular facilitation and passive vertebral mobilization for neck disability in patients with mechanical neck pain: A randomized controlled trial. J Bodyw Mov Ther. 2022 Jul;31:16-21. doi: 10.1016/j.jbmt.2022.02.009. Epub 2022 Mar 18. PMID 35710215